CLINICAL TRIAL: NCT04060888
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Ustekinumab in Chinese Subjects With Active Systemic Lupus Erythematosus
Brief Title: A Study of Ustekinumab in Chinese Participants With Active Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Pre-planned IA (global study) showed lack of efficacy in this indication. No new safety signals observed, findings consistent with known profile.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108631; CNTO1275SLE3003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ustekinumab (Experimental): Participants will receive ustekinumab approximately 6 milligram per kilogram (mg/kg) intravenously (IV) based on body weight-range at Week 0 followed by 90 mg ustekinumab subcutaneously (SC) at Week 8 and every 8 weeks (q8w) thereafter through Week 48 during double-blind period. Eligible participants who will enter the extension period will continue to receive 90 mg ustekinumab SC q8w through Week 160.
  Interventions: Drug: Ustekinumab (approximately 6 mg/kg); Drug: Ustekinumab 90 milligram (mg)
- Placebo (Placebo Comparator): Participants will receive matching placebo to ustekinumab IV at Week 0, followed by matching placebo to ustekinumab SC at Week 8 and q8w thereafter through Week 48 during double-blind period. Eligible participants who will enter the extension period will cross-over to receive 90 mg ustekinumab SC q8w through Week 160.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab (approximately 6 mg/kg) — Participants will receive ustekinumab approximately 6 milligram per kilogram via IV route based on body weight-range.
  Other Names: Stelara
  Arms: Ustekinumab
Drug: Ustekinumab 90 milligram (mg) — Participants will receive 90 mg ustekinumab via SC route.
  Other Names: Stelara
  Arms: Ustekinumab
Drug: Placebo — Participants will receive placebo matching to ustekinumab IV or SC.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab in Chinese participants with active systemic lupus erythematosus (SLE) who have not adequately responded to one or more standard-of-care treatments.

ELIGIBILITY:
Inclusion Criteria:

* Had a documented medical history (that is, met at least 1 of the two criteria below) that participant met the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for systemic lupus erythematosus (SLE) at least 3 months prior to first dose of study agent:

  1. Met a total of at least 4 SLICC criteria, including at least 1 clinical and at least 1 immunologic;
  2. Has a diagnosis of lupus nephritis, confirmed by renal biopsy and at least 1 of the following autoantibodies: antinuclear antibodies (ANA) or anti-double-stranded deoxyribonucleic acid (anti-dsDNA)
* Have a positive test in the medical history and confirmed at screening for at least 1 of the following autoantibodies: antinuclear antibodies, anti-double-stranded deoxyribonucleic acid, and/or anti-Smith
* Have at least 1 British Isles Lupus Assessment Group (BILAG) A and/or 2 BILAG B scores observed during screening
* Have a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score at least 4 (excluding diffuse non-inflammatory alopecia) or at least 4 joints with pain and signs of inflammation at screening, Week 0, or both
* Have a Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score greater than or equal to [>=] 6 at screening. Must also have SLEDAI-2K >= 4 for clinical features (excluding headache and laboratory abnormalities) at Week 0

Exclusion Criteria:

* Has any unstable or progressive SLE manifestation (example: central nervous system lupus, systemic vasculitis, end-stage renal disease, severe or rapidly progressive glomerulonephritis, pulmonary hemorrhage, myocarditis) that may warrant escalation in therapy beyond permitted background medications. Participants requiring renal hemodialysis or peritoneal dialysis are also excluded
* Has other inflammatory diseases that might confound the evaluations of efficacy (including but not limited to rheumatoid arthritis, psoriasis, psoriatic arthritis, Crohn's disease)
* Has urinary protein level of greater than (>) 4 gram per day (g/day) or protein/creatinine ratio estimating >4g/day equivalent proteinuria
* Has known allergies, hypersensitivity, or intolerance to ustekinumab or its excipients
* Has a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location, clinically significant splenomegaly, or history of monoclonal gammopathy of undetermined significance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-14 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index-4 (SRI-4) Composite Response at Week 52 | Week 52
  SRI-4 is a composite of at least 4 point improvement in Systemic Lupus Erythematosus Disease Activity Index 2000(SLEDAI-2K), no worsening in British Isles Lupus Assessment Group (BILAG) and no worsening in Physician's Global Assessment of Disease Activity score (PGA).

SECONDARY OUTCOMES:
Time to Flare | Baseline up to Week 52
  Time to flare is the duration of flare occurring at any time after the baseline will be calculated with flare defined as either 1 or more new British Isles Lupus Assessment Group (BILAG) A or 2 or more new BILAG B domain scores relative to baseline.
Percentage of Participants with an SRI-4 Composite Response at Week 24 | Week 24
  SLE Responder Index (SRI)-4 is a composite of at least 4 point improvement in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K, no worsening in BILAG and no worsening in PGA.
Percentage of Participants Achieving at Least a 50% Improvement in the Number of Joints with Pain and Signs of Inflammation at Week 52 | Week 52
  The percentage of participants achieving at least a 50 percent (%) improvement in the number of joints with pain and signs of inflammation at week 52 will be reported in participants with at least 4 affected joints at baseline.
Percentage of Participants Receiving Glucocorticoids at Baseline who Achieve Reduction in Glucocorticoid Dose by Week 40 and Sustain That Reduction Through Week 52 | Baseline up to Week 52
  Reduction of glucocorticoid dose is defined as a reduction in average daily oral glucocorticoid dose by at least 50% (relative to the baseline dose) or reduction of average daily oral glucocorticoid dose by at least 25% (relative to the baseline dose) so that the average daily dose is reduced to less than or equal to (<=) 7.5 milligram (mg) (prednisone or equivalent). Sustained reduction of glucocorticoid dose is defined as achieving an average daily oral glucocorticoid dose reduction between Weeks 24 and 40, and sustaining that reduction through Week 52, in those participants who, at baseline, were receiving oral glucocorticoids.
Percentage of Participants Achieving at Least a 50% Improvement in the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score at Week 52 | Week 52
  Percentage of participants achieving at least 50% improvement in CLASI Activity Score at Week 52 will be reported in participants with a CLASI Activity Score of 4 or greater at baseline.
Percentage of Participants Receiving Glucocorticoids at Baseline who Achieve Reduction in Glucocorticoid Dose by Week 40, Sustain That Reduction Through Week 52, and Achieve an SRI-4 Composite Response at Week 52 | Baseline up to Week 52
  Percentage of participants receiving glucocorticoids at baseline who achieve reduction in glucocorticoid dose by Week 40, sustain that reduction through Week 52, and achieve an SRI-4 composite response at Week 52 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069